CLINICAL TRIAL: NCT07124299
Title: Prospective, Randomized Study on the Efficiency of Alpha-Blockers Prior to Ureteral Sheath Placement in Flexible Ureterolithotripsy
Brief Title: Alpha-Blockers Prior to Ureteral Access Sheath Placement in Flexible Ureteroscopy: A Randomized Prospective Study
Acronym: ALFA-URS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Pedro de Figueiredo Buchalla (Other)
Responsible Party: Sponsor-Investigator, Pedro de Figueiredo Buchalla, Alpha-Blockers Prior to Ureteral Access Sheath Placement in Flexible Ureteroscopy: A Randomized Prospective Study, Centro Universitário FMABC
Organization: Centro Universitário FMABC (Other)
Allocation: Not Applicable | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMABC-ALFAURS-2025-01
Record Dates: First submitted 2025-08-09; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-05

CONDITIONS: Nephrolithiasis; Alpha Blocker; Ureteral Access Sheath
MeSH Terms: conditions — Nephrolithiasis | interventions — Observation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Alpha-blocker group (Active Comparator): Participants will receive an alpha-blocker (e.g., tamsulosin 0.4 mg orally once daily) for 7 consecutive days prior to flexible ureterorenolithotripsy. The medication aims to relax the ureteral smooth muscle and facilitate the insertion of the ureteral access sheath during surgery. All surgical procedures will follow the standard protocol used in the participating hospitals.
  Interventions: Drug: Experimental: Alpha-blocker group
- No Intervention: Control group (Placebo Comparator): Participants will undergo flexible ureterorenolithotripsy without the use of alpha-blockers prior to surgery. All other aspects of perioperative care and surgical technique will be identical to those of the experimental group.
  Interventions: Drug: No intervention (observational study)

INTERVENTIONS:
Drug: Experimental: Alpha-blocker group — Participants in the experimental arm will receive an oral alpha-blocker (tamsulosin 0.4 mg) once daily for 7 consecutive days before undergoing flexible ureterorenolithotripsy. The medication is intended to relax ureteral smooth muscle fibers, potentially facilitating the insertion of the ureteral access sheath and reducing the need for a secondary procedure. The dose, route, and timing are standardized for all participants in this arm.
  Arms: Experimental: Alpha-blocker group
Drug: No intervention (observational study) — Participants in this arm will undergo flexible ureterorenolithotripsy without receiving any alpha-blocker prior to surgery. All other perioperative care and surgical procedures will follow the same protocol as the experimental group.
  Arms: No Intervention: Control group

SUMMARY:
This study aims to evaluate whether the use of alpha-blockers before flexible ureterorenolithotripsy facilitates the passage of the ureteral access sheath. The trial will enroll adult patients diagnosed with kidney stones who are scheduled for flexible ureteroscopy. Participants will be randomly assigned to receive or not receive alpha-blockers for seven days before surgery. The primary outcome is the rate of successful sheath placement without the need for a second procedure. Secondary outcomes include the incidence of ureteral injuries and the need for additional surgical interventions. The goal is to improve surgical efficiency and patient outcomes in the treatment of kidney stones.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of nephrolithiasis with surgical indication for flexible ureterorenolithotripsy
* Ability to provide written informed consent

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* History of ureteral stricture, prior ureteral reconstructive surgery, and/or abdominal or pelvic radiotherapy
* Prior ureteroscopy or ipsilateral double-J stent placement within the past 3 months
* Chronic use of alpha-blockers for benign prostatic hyperplasia or medical expulsive therapy for ureteral stones

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in the failure rate of ureteral access sheath insertion with preoperative tamsulosin use | During the surgical procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Universitário FMABC, Santo André, São Paulo, Brazil